CLINICAL TRIAL: NCT03895788
Title: An Open-Label, Single-Arm, Phase I Clinical Trial to Evaluate the Safety and Tolerability of ZL-2306 (Niraparib) in Combination With Brivanib in Patients With Recurrent Ovarian Cancer
Brief Title: A Study of Niraparib in Combination With Brivanib in Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH1809001
Record Dates: First submitted 2019-02-28; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; brivanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- niraparib and brivanib (Experimental): Subjects will be assigned into niraparib 100mg+brivanib 200mg, niraparib 200mg+brivanib 200mg, niraparib 200mg+brivanib 400mg, niraparib 200mg+brivanib 600mg dose group at the first day of the first cycle.
  Interventions: Drug: niraparib; Drug: Brivanib

INTERVENTIONS:
Drug: niraparib — Niraparib will be administered as a flat-fixed dose (100mg or 200 mg, daily) depending on the cohort the patient is enrolled to, and not by body weight or body surface area. Each dose should be swallowed whole without chewing. The consumption of water is permissible. Patients should take doses at approximately the same times each day, and record this information in the patient diary. Patients will be provided with a diary in which to record their intake of study drug. However, the actual number of doses taken by the patient must be calculated from the number of tablets dispensed and returned.
Drug: Brivanib — Brivanib will be administered as a flat-fixed dose (200mg, 400 mg, or 600 mg daily) depending on the cohort the patient is enrolled to, and not by body weight or body surface area.

SUMMARY:
Open-label, cohort study to determine the safety and tolerability of the combination of daily niraparib and daily brivanib for one 28-day cycle in patients with advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent .
2. Female, age ≥ 18 years.
3. Histologically confirmed diagnosis of ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
4. Patients must have ovarian cancer and have failed at least 1 prior line of therapy
5. Life expectancy of more than 16 weeks.
6. ECOG 0-1.
7. Patient agrees to blood draws during study for the gBRCA test
8. Has good organ function, including:

   * Absolute neutrophil count ≥1,500/µL
   * Platelets ≥125,000/µL
   * Hemoglobin ≥10 g/dL
   * Serum creatinine ≤1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥60 mL/min using the Cockcroft-Gault equation
   * Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤1 x ULN
   * Aspartate aminotransferase and alanine aminotransferase ≤2.5 x ULN unless liver metastases are present, in which case they must be ≤5 x ULN
9. Female patient has a negative serum pregnancy test within 3 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 3 months after the last dose of study treatment, or is of non-childbearing potential. Non-childbearing potential is defined as follows (by other than medical reasons):

   * ≥45 years and <60 years of age and has not had menses for >1 year
   * ≥60 years of age
   * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation.
10. Is able to adhere to the protocol.
11. Has recovered from previous chemotherapy induced toxic side effects to ≤ grade 1 CTCAE or basal level, apart from ≤ grade 2 CTCAE peripheral neuropathy or hair loss symptoms at steady state.

Exclusion Criteria:

1. Has a known hypersensitivity to the active or inactive ingredients of ZL-2306 (niraparib) or compound which has similar chemical structure to ZL-2306 (niraparib).
2. Has a known hypersensitivity to the active or inactive ingredients of brivanib or compound which has similar chemical structure to brivanib.
3. Has symptomatic uncontrolled brain or leptomeningeal metastasis.
4. Major surgery or chemotherapy within 3 weeks of starting the study or patient has not recovered from any effects of the surgery.
5. Receive palliative radiotherapy encompassing > 20% of the bone marrow within 1 week of entering the study.
6. Be diagnosed any invasive cancer other than ovarian cancer (apart from cured basal cell carcinoma and squamous cell carcinoma) within 2 years prior to study enrolment.
7. Patient must has any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
8. Has other serious or uncontrolled disease
9. Has any disease, treatment and laboratory abnormality that may interfere the study results and affect the fully attendance of study. Or the patient is considered to be not suitable for the study by the investigator. Cannot receive platelet or red blood cell transfusion within 4 weeks of study drug administration.
10. Pregnant, breastfeeding or expecting to conceive children during the study treatment period.
11. Corrected QT (QTc) interval > 450 msec.
12. Prior PARP inhibitor therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 1 year
  To determine the maximum tolerated dose of the combination of niraparib and brivanib for the treatment of patients with advanced ovarian cancer. The maximum tolerated dose (MTD) that is defined as the dose level at which less than one-third of patients will experience a dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Assess the toxicity of the combination of niraparib and brivanib in each cohort by number of participants with treatment related adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Jing Wang, Changsha, Hunan, China